CLINICAL TRIAL: NCT04650945
Title: In-hospital Diabetes Management With Flash Glucose Monitoring (isCGM) - the INDIGO Study, Part A
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staff shortage
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Julie Støy, Principal investigator, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1-10-72-188-20
Record Dates: First submitted 2020-11-13; First posted 2020-12-03 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus; Diabetes Mellitus
Keywords: Continuous glucose monitoring; Hospitalization; Nutritional therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- isCGM-arm (Active Comparator): isCGM (intermittently scanned continuous glucose monitor) data obtained from a FreeStyle Libre Flash continuous glucose monitoring system will be viewed real-time and used to adjust diabetes treatment
  Interventions: Other: isCGM group
- POC-arm (No Intervention): POC glucose readings are used to adjust diabetes treatment. CGM data from the Freestyle Libre monitor are blinded to all and only gathered for comparison purposes to intervention group.

INTERVENTIONS:
Other: isCGM group — As previously described
  Arms: isCGM-arm

SUMMARY:
The aim of the study is to investigate the applicability of a Flash glucose monitoring sensor (Freestyle Libre, isCGM) for in-hospital glucose monitoring in patients with diabetes requiring nutritional therapy (tube feeding or parenteral feeding).

DETAILED DESCRIPTION:
All patients who meet study criteria will be invited to participate in the study. All patients included in the study will be followed by a trained clinical diabetes specialist and a trained study nurse (study personnel) for glucose management during their hospitalization. All patients included in the study will receive a Freestyle Libre isCGM. The patients will be randomized to control (blinded isCGM glucose values to patient and study personnel and POC (point-of-care) plasma glucose will be used for adjusting diabetes treatment) or intervention (isCGM blood glucose values will be used to aid with glucose management during the hospitalization). The study personnel will work with the patient's care team.

ELIGIBILITY:
Inclusion Criteria:

* Expected length of hospital stay of at least 48 hours
* Diagnosed with diabetes
* Literate in Danish
* Nutritional therapy using tube feeding or parenteral nutritional therapy
* Admission to Department of Gastrointestinal Surgery or Department of Heart-, Lung-, and Vascular surgery, both at Aarhus University Hospital, Denmark.

Exclusion Criteria:

* Pregnancy
* Patient unable to provide informed consent
* Patient unable to use mobile phone for reading isCGM sensor
* Known allergy to adhesives
* Anticipated MRI during the hospital admission
* Patients using CGM prior to hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Glucose time in range (3,9-10 mmol/l) (% pr day) | 2-14 days
  Glucose time in range (3,9-10 mmol/l) when diabetes treatment is adjusted using isCGM compared with standard care using POC plasma glucose monitoring (PG) (% pr day)

SECONDARY OUTCOMES:
Mean glucose (mmol/l) isCGM versus POC PG | 2-14 days
  Mean glucose (mmol/l) when diabetes treatment is adjusted using isCGM compared with standard care using POC plasma glucose monitoring (PG)
Glycemic variability; coefficient of variation (CV) (in %) | 2-14 days
  CV when diabetes treatment is adjusted using isCGM compared with standard care using POC plasma glucose monitoring (PG)
Glycemic variability; standard deviation (SD) | 2-14 days
  SD when diabetes treatment is adjusted using isCGM compared with standard care using POC plasma glucose monitoring (PG)
Time in hypoglycemia (<3 mmol/L) (%) | 2-14 days
  Time in hypoglycemia (%) when diabetes treatment is adjusted using isCGM compared with standard care using POC plasma glucose monitoring (PG)
Time in hypoglycemia (<3,9 mmol/l) (%) | 2-14 days
  Time in hypoglycemia (%) when diabetes treatment is adjusted using isCGM compared with standard care using POC plasma glucose monitoring (PG)
Number of events with hypoglycemia (<3,9 mmol/l) (%) | 2-14 days
  Number of events with hypoglycemia per day (<3,9 mmol/L for >15 minutes) when diabetes treatment is adjusted using isCGM compared with standard care using POC plasma glucose monitoring (PG)
Time in hyperglycemia (>10 mmol/l) (%) | 2-14 days
  Time in hyperglycemia when diabetes treatment is adjusted using isCGM compared with standard care using POC plasma glucose monitoring (PG)
Glucose out of range: Time in hypoglycemia and time in hyperglycemia (<3,9 and >10 mmol/l) (%) | 2-14 days
  Glucose out of range: Time in hypoglycemia and time in hyperglycemia (<3,9 and >10 mmol/l) (%) when diabetes treatment is adjusted using isCGM compared with standard care using POC plasma glucose monitoring (PG)
Daily total insulin dosage (IE) | 2-14 days
  Daily total insulin dosage (IE) when diabetes treatment is adjusted using isCGM compared with standard care using POC plasma glucose monitoring (PG)
Time with active isCGM | 2-14 days
  Time with active isCGM (%) in intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Julie Støy, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus university hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No